CLINICAL TRIAL: NCT03252197
Title: A Randomized Parallel Study for Simulated Internal Jugular Vein Cannulation Using Simple Needle Guide Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2016-0081
Record Dates: First submitted 2017-07-28; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Doctors Attending a Central Line Insertion Training Courses for New Residents of a University Hospital From March 2017 to June 2017; Physicians Who Had Less Than 10 Ultrasound Guided Internal Jugular Vein Cannulation Participate in This Study
Keywords: Ultrasound guided central venous cannulation; new device; first attempt success

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded to study arm, Outcome assessor measured outcome variables based on recorded images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New device group (Experimental): participants who are tested performance for ultrasound guided cannulation using device
  Interventions: Device: UGIJVC with needle guide device
- Conventional group (Active Comparator): participants who are tested performance for ultrasound guided cannulation using conventional method
  Interventions: Device: UGIJVC without needle guide device

INTERVENTIONS:
Device: UGIJVC with needle guide device — Study subjects assigned to each group were trained in ultrasound guided internal jugular venous cannulation (UGIJVC) in separate spaces. On each session, subjects were educated about UGIJVC for 30 minutes, and the instructor who was in charge of session, consisted of experienced physicians who had 50 or more UGIJVC success experiences without a supervisor in clinical field. The instructors explained the anatomical structure and the principles of UGIJVC and then demonstrated the procedures directly to the subjects using phantom. After that, all subjects were instructed to perform hands on practice for 30 minutes. In case group, the instructor trained subjects using device. On the other hand in control group, UGIVJC was demonstrated as a conventional method of approaching the target vessel while confirming the needle tip on the ultrasound screen in real time without a device.
  Arms: New device group
Device: UGIJVC without needle guide device — participants who are tested performance for ultrasound guided cannulation using conventional method.
  Other Names: Conventional group
  Arms: Conventional group

SUMMARY:
Two-dimensional ultrasound guided approach does not guarantee first attempt success on internal jugular vein cannulation. New attachable device recently was developed for accurate needle insertion when ultrasound is used. Our randomized parallel simulation study will examine whether this device will improve the first attempt success rate when ultrasound guided internal jugular vein catheterization of simulated internal jugular vein.

DETAILED DESCRIPTION:
This was a prospective, randomized, parallel trial using phantom simulating internal jugular vein.

After informed consent all subjects will be randomized to insert needle for internal jugular vein cannulation of phantom using ultrasound approach with or without this device. Video camera will record all procedure process and ultrasound image in real time. Researchers blinded to the study aim measured outcome variables based on recorded images.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 20
2. Resident in clinical hospital
3. Ultrasound-guided internal jugular vein insertion without supervisor experience less than 10

Exclusion Criteria:

1. If they have physical problem that is difficult to perform
2. If they do not want to participate in this study
3. If they can not understand the contents reading the informed consent
4. If they have more than 10 ultrasound guided internal jugular vein insertion without supervisor

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-03-11 (Actual); Primary Completion 2017-06-24 (Actual); Study Completion 2017-06-24 (Actual)

PRIMARY OUTCOMES:
First attempt success | Within 2 minutes or after start to insertion attempt
  The first attempt success was defined as a successful attempt to perform a vein puncture in one attempt. The number of attempts was counted each time a subject inserted a guide needle into the phantom surface, followed by withdrawal, redirect, or reinsertion.

SECONDARY OUTCOMES:
Posterior wall puncture of the internal jugular procedure, comfort level with procedure | Within 2 minutes or after start to insertion attempt
  It was defined when the needle tip on the recorded ultrasound screen was confirmed to pass through the posterior wall measurement unit : Yes or no (categorical variable)
Carotid artery puncture | Within 2 minutes or after start to insertion attempt
  It was defined as the needle tip passing through the carotid lumen or the subject regurgitating artery water during cannulation attempt.
  measurement unit : Yes or no (categorical variable)
Time to cannulation | Within 2 minutes or after start to insertion attempt
  It was defined as the time from time out for procedure start to end point measurement unit : second
Comfort level | Within 2 minutes or after start to insertion attempt
  It was defined subjective opinion about difficulty during procedure for each subject measurement unit : 100-mm visual analogue scale with 0 being the least of the difficulties and 10 being the highest.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Yonsei University College of Medicine, Yonsei University Severance Hospital, Seoul, South Korea